CLINICAL TRIAL: NCT02766192
Title: Ketamine and Mindfulness Based Cognitive Therapy (MBCT) in Treatment of Post-Traumatic Stress Disorder (PTSD): Comparison of Treatment Efficacy and Metabolomic Profiles
Brief Title: TIMBER Psychotherapy and Ketamine Single Infusion in Chronic PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-078
Record Dates: First submitted 2016-04-11; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: PTSD
Keywords: ketamine; mindfulness based cognitive therapy; PTSD; trauma memory; memory extinction; memory re-consolidation; metabolomics; TIMBER (Trauma Intervention using Mindfulness Based Extinction and Re-consolidation of trauma memories)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TIMBER-Ketamine arm (Experimental): This arm received TIMBER psychotherapy and ketamine infusion.
  Interventions: Drug: Ketamine; Behavioral: TIMBER Psychotherapy
- TIMBER-placebo arm (Placebo Comparator): This arm received TIMBER psychotherapy and placebo (normal saline) infusion.
  Interventions: Behavioral: TIMBER Psychotherapy; Drug: Placebo (normal saline)

INTERVENTIONS:
Drug: Ketamine
  Arms: TIMBER-Ketamine arm
Behavioral: TIMBER Psychotherapy
Drug: Placebo (normal saline)
  Arms: TIMBER-placebo arm

SUMMARY:
Background: The poor prognosis and public health burden of PTSD necessitates the development of more effective and broader treatment approaches. In the etiopathogenesis of PTSD, trauma memories become ingrained into key brain areas through conditioned learning and are triggered by various situations of daily life. The brain glutamate system plays a key role in the process of trauma learning and trauma memories via long-term potentiation. Ketamine administration modulates the glutamate system and has been used in the treatment of depression and PTSD. Previous studies demonstrate that a single low dose of ketamine rapidly improves symptoms of refractory PTSD and treatment resistant depression. Unfortunately the observed response is short-lived (4-7 days, maximum up to 2 weeks) and multiple doses often produce unacceptable side effects. TIMBER (Trauma Interventions using Mindfulness Based Extinction and Reconsolidation for trauma memory) psychotherapy, is a manualized and translational mindfulness based cognitive behavioral therapy specifically designed to target trauma memories and their expressions in PTSD patients. The placebo controlled pilot study examined the efficacy of a protocol combining a single infusion of low dose ketamine (0.5mg/kg) and TIMBER psychotherapy in subjects suffering from chronic PTSD. The objective of this pilot study was to optimize and individualize treatment of chronic PTSD using a rapid, effective, trauma specific, user friendly and inexpensive approach that uses cutting edge psychopharmacological combined with novel psychotherapeutic approaches.

Methodology: The randomized, double blind, placebo-controlled pilot study used a crossover design. Ten subjects with refractory PTSD were assigned to one of two arms: one arm (n=5) received combined ketamine infusion and TIMBER therapy (TIMBER-K arm) and the second (n=5) received combined placebo (normal saline) infusion and TIMBER therapy (TIMBER-P arm). All 10 subjects received a short version of TIMBER therapy after 10 minutes of onset of the infusion in which reactivation of trauma memories was initiated in a controlled manner using standardized scales and scripted narrative of the index trauma. This was followed by a standardized mindfulness based cognitive therapy module to quickly de-escalate the arousal symptoms followed by induction of detached observation and reappraisal of the trauma experience. After completion of the 40-min infusion, all subjects were trained on the full version of TIMBER therapy using methods of mindfulness based graded exposure therapy and a twice-daily schedule of home practice was initiated. The investigators are currently in a process of recruiting fifty more subjects to examine the effects in a larger sample.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, 21-60 years of age;
2. Patients attending the outpatient psychiatry clinic of Cooper University Hospital will be screened for this study using DSM-IV diagnostic criteria for PTSD.
3. Participants must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign a written informed consent document;
4. Participants must fulfill DSM-IV criteria for current civilian or combat-related PTSD, based on clinical assessment by a study psychiatrist, on the self-rated PTSD Check list (PCL-C scores must be at least 51and CAPS score must be at least 50 at screening on the first 17 items of the scale).
5. Women must be using a medically accepted reliable means of contraception (oral contraceptive medication etc.) or not be of childbearing potential (i.e., surgically sterile, postmenopausal for at least one year);
6. Women of childbearing potential must have a negative pregnancy test at screening and pre-infusion;
7. Throughout this study, the participants will be on stable dosage(s) of medication(s).

Exclusion Criteria:

1. Meet criteria for psychotic disorders, e.g. schizophrenia/ schizoaffective disorder.
2. Women who are pregnant or are breast-feeding (because the medical risk of using ketamine during pregnancy and breast-feeding are unknown);
3. Serious, unstable medical illnesses such as hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease (including obstructive sleep apnea, history of difficulty with airway management during previous anesthetics, ischemic heart disease and uncontrolled hypertension, and history of severe head injury);
4. Clinically significant abnormal findings of laboratory parameters, or physical examination;
5. Patients with uncorrected hypothyroidism or hyperthyroidism;
6. Histories of mental retardation
7. History of one or more seizures without a clear and resolved etiology;
8. Drug or alcohol abuse or dependence within the preceding 3 months: phencyclidine (PCP) is especially important in this context because of its resemblance with ketamine not only in structure but also its pharmacodynamic effects on NMDA receptors.
9. Previous recreational use of ketamine;
10. Diagnosis of schizotypal or antisocial personality disorder (since these are known to reduce the possibility of study completion; other Axis II diagnoses will be allowed).

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-08; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline scores on the Clinician Administered PTSD Scale (CAPS) at 25th hours post-infusion | For CAPS, change in scores at 25th hour post-infusion compared to the baseline were measured
  Response (or Relapse status) was assessed by determining the change from baseline scores on the Clinician Administered PTSD Scale (CAPS) at Days-1 (25th hour post-infusion), 7, 14, 21, 28, 35, 42 and 49 and so on following the initiation of the protocol. This was done in this weekly fashion till 3 months after the infusion. A subject was considered to have relapsed when his/her scores were >50 in the CAPS scale and >51 in PTSD Symptom Checklist (PCL) scale respectively. A subject was considered to be a 'Responder' when there was a reduction of 20 or more points of these scores at 25th hours post-infusion compared to his/her baseline scores on CAPS and PCL. To be considered a responder, the response needed to be sustained for 7 days or more.
Change from baseline scores on the PTSD Symptom Checklist (PCL, self-reported) at 25th hours post-infusion | For PCL, change in scores at 25th hour post-infusion compared to the baseline were measured
  Response (or Relapse status) was assessed by determining the change from baseline scores on the PTSD Symptom Checklist (PCL) at Days-1 (25th hour post-infusion), 7, 14, 21, 28, 35, 42 and 49 and so on following the initiation of the protocol. This was done in this weekly fashion till 3 months after the infusion.
  Both CAPS and PCL scales are used in this study to ensure accuracy and objectivity.

SECONDARY OUTCOMES:
Change from baseline scores on the Hamilton depression rating scale (17-item version) at 25th hours post-infusion | For Hamilton depression rating scale, change in scores at 25th hour post-infusion compared to the baseline were measured
Change from baseline scores on the Beck Anxiety Scale at 25th hours post-infusion | For Beck Anxiety Scale, change in scores at 25th hour post-infusion compared to the baseline were measured

CONTACTS AND LOCATIONS:
Overall Officials: Basant Pradhan, MD, Principal Investigator — Cooper Health System
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pradhan B, Kluewer D'Amico J, Makani R, Parikh T. Nonconventional interventions for chronic post-traumatic stress disorder: Ketamine, repetitive trans-cranial magnetic stimulation (rTMS), and alternative approaches. J Trauma Dissociation. 2016;17(1):35-54. doi: 10.1080/15299732.2015.1046101. Epub 2015 Jul 10. PMID 26162001
- [Result] Pradhan B, Parikh T, Makani R, Sahoo M. Ketamine, Transcranial Magnetic Stimulation, and Depression Specific Yoga and Mindfulness Based Cognitive Therapy in Management of Treatment Resistant Depression: Review and Some Data on Efficacy. Depress Res Treat. 2015;2015:842817. doi: 10.1155/2015/842817. Epub 2015 Oct 5. PMID 26509083
- See also: Depression Specific Yoga and Mindfulness Based Cognitive Therapy in Management of Treatment Resistant Depression: Review and Some Data on Efficacy. — http://www.ncbi.nlm.nih.gov/pubmed/?term=26509083